CLINICAL TRIAL: NCT07345221
Title: Effect of Hilotherapy on Quality of Life and Comfort Level in the Management of Symptoms Related to Taxane-Associated Peripheral Neuropathy in Breast Cancer Patients
Brief Title: Effect of Hilotherapy in the Management of Symptoms Related to Taxane-Associated Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuran Ayşen Pamir Aksoy (Other)
Responsible Party: Sponsor-Investigator, Nuran Ayşen Pamir Aksoy, Assist. Prof., Acibadem University
Organization: Acibadem University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-13-470
Record Dates: First submitted 2025-06-04; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Peripheric Neuropathy
Keywords: hilotherapy; peripheric neuropathy; symptom management; pain; comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Hilotherapy
  Interventions: Device: Hilotherapy
- Control group (No Intervention): Non-hilotherapy

INTERVENTIONS:
Device: Hilotherapy — Applying hilotherapy device at chemotherapy courses
  Arms: Study Group

SUMMARY:
In this randomized controlled study, it was aimed to determine the effect of hilotherapy on quality of life and comfort level in the management of symptoms related to taxane-associated peripheral neuropathy in patients with breast cancer.

* The experimental and control group patients will answer the survey questions according to the data collection forms before the first chemotherapy course (To) and will undergo physical examinations by the researcher.
* In the experimental group, the Hilotherapy device will be connected and initiated 30 min before the chemotherap.
* The device will continue to cool for another 60 minutes when the chemotherapy ends.
* Both groups will continue to receive chemotherapy courses at the intervals determined as planned.
* Hilotherapy will be applied to the experimental group patients during each course according to the study protocol.
* For both groups, participants will answer the questions according to the data collection forms and will undergo physical examinations by the researcher after the 4th chemotherapy course (T1), 8th chemotherapy course (T2), 12th chemotherapy course (T3) and 4 weeks after the end of chemotherapy (T4).

DETAILED DESCRIPTION:
Hilotherapy Device Usage

1. 30 minutes before chemotherapy, disposable cellulose covers are placed on the patient's clean hands and feet (for hygiene and to prevent contamination)
2. The device is set to 12°C for hands and 14°C for feet.
3. Sensors are monitored during chemotherapy.
4. The hylotherapy application is continued for another 60 minutes after the end of the chemotherapy course.
5. At the end of the period, the sleeves and disposable covers are removed.

Data Collection Tools of the Study

* Introductory Information Form (designed by the researchers)
* "Other Methods Used by the Patient to Prevent Peripheral Neuropathy" Form
* Hilotherapy Application Data Form
* LANSS Pain Scale
* European Organization for Research and Treatment of Cancer Quality of Life Scale (EORTC QLQ-C30)
* European Organization for Research and Treatment of Cancer Quality of Life Chemotherapy-Associated Peripheral Neuropathy Scale (EORTC QLQ-CIPN20)
* General Comfort Scale-Short Form

ELIGIBILITY:
Inclusion Criteria:

* Having a primary breast cancer diagnosis
* Having received chemotherapy containing taxane compounds due to breast cancer
* Not having been previously diagnosed with peripheral neuropathy

Exclusion Criteria:

* Presence of distant metastasis
* History of psychiatric disorder
* Diagnosed diseases such as diabetes mellitus, autoimmune disease, megaloblastic anemia, cervical/spinal disc herniation, Raynaud's
* Active lesions on hands or feet
* Bleeding/clotting disorder
* Extremity amputation
* Any problem that prevents cognitive, emotional and verbal communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Taxan-induced peripheric neuropathy score | Will be assessed at the following time points: • Baseline -Week 0 (before chemo) • Week 4 (end of 4th chemo cycle) • Week 8 (end of 8th chemo cycle) • Week 12 (end of 12th chemotherapy cycle; last treatment) • Week 16 (4 weeks after completion of chemo)
  Taxan-induced peripheric neuropathy score measured by "European Organization for Research and Treatment of Cancer Quality of Life Chemotherapy-Related Peripheral Neuropathy Scale (EORTC QLQ-CIPN20)" The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy 20-item scale (EORTC QLQ-CIPN20) is a specific tool for determining TIPN symptoms. This patient-reported questionnaire comprises 20 items that can be divided into 3 subscales (sensory-9 items, motor-8 items, and autonomic-2 items. Item 39 is not included in any subscale and is analyzed separately as a single item). Responses follow a 4-point Likert scale:
  1. = "Not at all"
  2. = "A little"
  3. = "Quite a bit"
  4. = "Very much" Interpretation Higher total scores (closer to 100) = More severe neuropathy symptoms Lower total scores (closer to 0) = Fewer/milder symptoms

OTHER OUTCOMES:
General comfort level of patients | Will be assessed at the following time points: • Baseline -Week 0 (before chemo) • Week 4 (end of 4th chemo cycle) • Week 8 (end of 8th chemo cycle) • Week 12 (end of 12th chemotherapy cycle; last treatment) • Week 16 (4 weeks after completion of chemo)
  Confort level assessed by "General Comfort Scale Short Form". Is is a condensed version of the original Kolcaba General Comfort Questionnaire, designed to assess a patient's comfort levels across physical, psychospiritual, environmental, and sociocultural domains. The short form includes 28 items and uses a 6-point Likert scale. (1 = Strongly Disagree (least comfort) - 6 = Strongly Agree (most comfort)) Interpretation Higher scores (↑) = Better comfort (e.g., 70-100 = high comfort). Lower scores (↓) = Discomfort or unmet needs (e.g., <50 = significant discomfort).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acibadem Altunizade Hospital, Istanbul
  - Acibadem Maslak Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided